CLINICAL TRIAL: NCT04286269
Title: Effects of Music Based Intervention (MBI) on Pain Response and Neurodevelopment in Preterm Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid constraints on recruitment
Sponsor: University of Minnesota (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEUR-2019-27528; 1R61AT010712-01 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Preterm Birth; Pain
Keywords: Music Based Intervention; Preterm Infant Pain Profile
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be maintained by using identical headphones and MP3 players for all subjects. The PI, any personnel involved in collecting the clinical outcomes (e.g., PIPP) or collecting or quantifying EEG outcomes, and the statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this group will be randomized to receive the intervention.
  Interventions: Other: Music Based Intervention
- Placebo (Sham Comparator): Participants in this group will be randomized to receive a sham treatment.
  Interventions: Other: Sham Treatment

INTERVENTIONS:
Other: Music Based Intervention — Participants assigned to MBI will receive a total of 1.5 hours of music intervention 5-6 sessions per week. Music will be alternating: 30 minutes on and 30 minutes off and will be played when the subject is awake to cue pacification and initiate the sleep process. Music will be delivered through headphones using an MP3 player.
  Arms: Intervention
Other: Sham Treatment — Participants assigned to the control group will have the same treatment as the MBI group, but with no sound played through the headphones.
  Arms: Placebo

SUMMARY:
Pilot prospective randomized, double blinded, controlled study to test effect of music based intervention (MBI) on pain response and neurodevelopment in preterm infants.

DETAILED DESCRIPTION:
Aim 1: Premature infant pain profiles (PIPP) include physiologic, behavioral, and contextual measures which identifies differences in pain responses between music-based intervention (MBI) and controls while still in the neonatal intensive care unit (NICU). Central EEG amplitude changes have been time-locked with painful procedures in term infants. We will explore if PIPP scores and central EEG amplitude changes are attenuated with MBI in comparison to controls.

Hypothesis 1: MBI will show improved pain responses, with lower PIPP scores and attenuated central EEG amplitude changes during painful procedures, in comparison to the control cohort.

Aim 2: EEG is a surrogate marker for real time brain function during sleep-wake cycles. Because preterm brain networks develop during sleep, sleep duration is a strong indicator of brain maturation. Serial biweekly EEGs of preterm infants can quantify sleep duration trends and track MBI's influence on sleep. To enhance objectivity, innovative EEG machine-learning tools will be applied to the analyses.

Hypothesis 2: MBI will enhance preterm EEG brain maturation in comparison to controls.

Due to the natural limitations of evaluating immature neonatal nervous systems, ERPs have been utilized to study early neurodevelopment. ERPs quantify electrical brain potentials changes time-locked with a stimulus. Auditory ERPs performed at 1 month corrected age evaluates attention and discrimination between familiar and novel stimuli - early neurodevelopmental signs of recognition memory function and perceptual learning.

Hypothesis 3: ERPs at 1 month corrected age will show that MBI has a greater impact on early neurodevelopment when compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant born at 30 weeks (+/- 2 weeks)
* Medically stable

Exclusion Criteria:

* Treatment for major organ system disease
* Significant neurological disorder including, but not limited to, abnormal neurological examination, neonatal abstinence syndrome, intraventricular hemorrhage, seizures, meningitis, or congenital brain malformations
* Scalp lesions affecting EEG placement

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Wang, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 14 | 14
Completed | 7 | 9
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 28
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Premature Infant Pain Profile (PIPP) Score
Description: The Premature Infant Pain Profile (PIPP) is a pain scoring system assessing 7 indicators: observed change in heart rate, observed decrease in percent oxygen saturation; observed facial expressions of pain (brow bulge, eye squeeze, and naso-labial furrow); gestational age; and behavioral state. Clinicians rate each indicator on a scale from 0 to 3 using a set scoring system. Total scores range 0 to 21, with higher scores indicating greater pain.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: unit in a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 10 | 13
unit in a scale | 6.8 (3.6) | 7.8 (3.7)

2. Primary Outcome: Premature Infant Pain Profile (PIPP) Score
Description: as for outcome 1
Time Frame: 4 weeks
Population: .All other outcome measures besides 1 were considered separate. Each outcome measure had a different number of participants who completed that portion of the study. The ERP (Event Related Potential) measure only had one participant attend. Ultimately, the number of participants analyzed should be based on the first primary outcome measure of pain profile.
Measure: Mean (Standard Deviation); unit: unit in a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 7 | 9
unit in a scale | 6.3 (2.7) | 6.4 (3.5)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Description: Adverse events not collected
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT04286269/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT04286269/ICF_001.pdf